CLINICAL TRIAL: NCT01435252
Title: A Phase II, Randomized, Open-Label, Single Center Study In Patients With Advanced Head And Neck Cancer To Investigate Efficacy And Safety Of Standard Chemoradiation And Add-On Concurrent Cetuximab ± Consolidation Cetuximab
Brief Title: A Phase II Study In Patients With Advanced Head And Neck Cancer Of Standard Chemoradiation And Add-On Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Oliver Riesterer, Leitender Arzt, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Add-On cetuximab
Record Dates: First submitted 2011-07-26; First posted 2011-09-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Oropharyngeal Cancer; Hypopharyngeal Cancer; Laryngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients will be treated with chemoradiation in combination with concurrent cetuximab. Two weeks after end of chemoradiation the consolidation phase will start and patients will receive biweekly consolidation cetuximab, maximally 6 infusions over 12 weeks.
  Interventions: Drug: Cetuximab
- Arm B (Experimental): Patients will be treated with chemoradiation in combination with concurrent cetuximab.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Arm A: chemoradiation in combination with concurrent cetuximab Arm B: chemoradiation in combination with concurrent and consolidation cetuximab
  Other Names: Erbitux®

SUMMARY:
Sixty patients with advanced squamous cell carcinomas of the head and neck will be enrolled in this study. Patients are treated with standard chemoradiation in combination with concurrent add-on cetuximab. Subsequently patients are randomized to cetuximab consolidation therapy (three months, Arm A) versus no consolidation therapy (Arm B). The aim of this study is to investigate if cetuximab consolidation therapy improves the 2-year locoregional control rate.

* Trial with medicinal product
* Trial with radiotherapy

DETAILED DESCRIPTION:
This clinical study translates our preclinical findings that concurrent and consolidation cetuximab improves efficacy of RT into the clinic. It is a phase II, randomized, open-label, single center study in patients with locoregionally advanced stage III-IV and/or total gross tumor volume (tGTV) > 70cc head and neck cancer. This study population is at high risk for locoregional recurrence after chemoradiation alone. Tumor stages to be included are T3-4 Nx, Tx N2b-N3 (N2b only if ≥ 3 ipsilateral nodes involved) M0 and/or tGTV >70 cc (any T, any N, M0) squamous cell cancers of the head and neck (HNSCC). All patients will receive in, the so called 'Induction Phase' standard chemoradiation (RT up to 70 Gy in combination with weekly CDDP 40 mg/m2) and add-on concurrent cetuximab (loading Dose 400 mg/m2, concurrent dose 250 mg/m2 weekly). The patients are randomized to either add-on consolidation cetuximab (500 mg/m2 biweekly x 6 over 12 weeks) (Arm A) or no further treatment (Arm B). Randomization will take place after Induction Phase. The total number of patients to be included into the study is 60 (30 patients per arm). Up to 6 patients may be replaced in case of early drop out to reach that aim.

The sample size of 60 patients is considered to be sufficient to collect first information on clinical efficacy and the possible impact of various biomarkers on clinical endpoints. If the results of this study will demonstrate that the novel treatment regimen is safe and efficacious, a randomized multicenter phase III study will follow.

ELIGIBILITY:
Inclusion criteria:

* T3-4 Nx M0; Tx N2b-3 M0 (N2b only if ≥ 3 ipsilateral nodes involved) and/or total GTV > 70 cc (any T, any N, M0)
* biopsy proven squamous cell cancer
* primary tumor location in oral cavity, oropharynx, hypopharynx or larynx
* Patients with CUP (cancer of unknown primary) syndrome in case they have advanced lymph node metastases (Tx N2b-3 M0 (N2b only if ≥ 3 ipsilateral nodes involved).- Indication for chemoradiation (RT + Cisplatin)
* curative treatment intent
* Start of chemoradiation within the recruitment time frame
* Performance Status WHO/ECOG: 0-1
* Age between 18 and 75 years
* No previous chemotherapy or RT for cancer of the head and neck
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study (until at least 60 days following the last study treatment
* Patient must sign informed consent prior to study entry.

Exclusion criteria:

* Cancer of the nasopharynx
* Any neoadjuvant chemotherapy prior to screening
* Treatment with other investigational drugs within 4 weeks
* History of malignancy other than basal cell skin cancer unless disease free for a minimum of 3 years.
* Uncontrolled claudication, bleeding, or thromboembolic disorders at screening
* Patients receiving heparin, warfarin or phenprocoumon therapy are ineligible- Uncontrolled and severe hypertension at screening according to the judgement of the investigator.
* Current uncontrolled cardiac disease: Unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, history of myocardial infarction within 12 months, significant arrhythmias
* Left ventricular function < 45 % (determination of left ventricular function required when history of cardiac disease)
* History of stroke within 6 months
* Major surgical procedure, or significant traumatic injury within 28 days prior to screening; anticipation of need for major surgical procedure during the course of the study.
* Acute bacterial or fungal infection requiring intravenous antibiotics at screening
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at screening
* Pregnant (positive pregnancy test) or lactating
* Previous organ transplantation
* Any immune suppressive therapy
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition because study treatment might be immuno-suppressive (Note: HIV testing only required if clinically indicated)
* Any uncontrolled condition, which in the opinion of the investigator, would interfere with the safe and timely completion of study procedures.
* Preexisting renal insufficiency with impaired creatinine clearance (<60ml/min) and/or increased plasma creatinine (>106 µmol/l) at screening
* History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to screening
* Serious, non-healing wound, ulcer, or bone fracture
* AST, ALT, or bilirubin > 1.5 x normal
* Preexisting absolute neutrophil count (ANC) < 1,800 cells/mm3
* Platelets < 100,000 103/µl at screening
* PTT > 1.5 x normal
* WBC < 4000 103/µl
* Hb < 11 g/dl at screening (Note: The use of transfusion or other intervention to achieve Hb > 11 g/dl is possible)
* Contraindication to CDDP
* Known allergy to cetuximab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Locoregional tumor control | 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Metastasis rate | 2 years
Metastasis free survival (MFS) | 2 years
Biological surrogate markers | 2 years
Safety and tolerability | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Riesterer, Leitender Arzt, Principal Investigator — University Hospital Zurich, Division of Radiation Oncology
Locations (1):
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] de Galiza Barbosa F, Riesterer O, Tanadini-Lang S, Stieb S, Studer G, Pruschy M, Huber GF, Huellner MW, Stolzmann P, Veit-Haibach P. Evaluation of 18F-FDG PET/CT as an early imaging biomarker for response monitoring after radiochemotherapy using cetuximab in head and heck squamous cell carcinoma. Head Neck. 2020 Feb;42(2):163-170. doi: 10.1002/hed.25975. Epub 2019 Nov 9. PMID 31705729